CLINICAL TRIAL: NCT02886975
Title: Effects of Low Protein Diet Supplemented Keto-/Amino Acid in Preventing the Progression of Chronic Kidney Disease(CKD)
Brief Title: Effects of Low Protein Diet in Preventing the Progression of Chronic Kidney Disease(CKD)---a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YYK-2016001
Record Dates: First submitted 2016-08-07; First posted 2016-09-01 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Renal Insufficiency, Chronic; Diet, Protein-Restricted
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- low protein diet plus α-keto acid (Experimental): A comparison of normal diet and low protein diet plus α-keto acid after intervention in the same individual
  Interventions: Behavioral: low protein diet plus α-keto acid

INTERVENTIONS:
Behavioral: low protein diet plus α-keto acid — 0.4-0.6g of proteins per kilo of body weight per day, supplemented with α-keto acid tablets
  Other Names: low protein diet

SUMMARY:
The purpose of this study is to determine whether low protein diet and very low protein diet supplemented keto-/amino acid is effective in preventing the progression of chronic kidney disease (CKD , stage 2 to 5).

DETAILED DESCRIPTION:
Dietary protein restriction represents a basic therapeutic approach in chronic kidney disease(CKD), by reducing the accumulation of nitrogen catabolic substances, and by delaying the progress of CKD and proteinuria, but the effects of the low protein diet on renal failure progression rate remain to be determined.The aim of this study is to evaluate the efficacy of low protein diet and α-keto acid tablet in retard the progress of CKD. This is a prospective study, 100 patients who meet inclusion and exclusion criteria will be included. The changes of glomerular filtration rate in CKD and time to renal replacement will be evaluated after 1 year treatment.

ELIGIBILITY:
Inclusion Criteria: Patients with chronic kidney disease in stage 2 to 5 (GFR<60 ml/min/1.73m2) receiving conservative treatment for CKD

Exclusion Criteria: None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
changes in glomerular filtration rate | 1 year
  Nutritional status, evaluated by nutrition risk screening (NRS 2002), at the start and during the 1st year of investigators' intervention.

SECONDARY OUTCOMES:
Compliance to diet | 1 year
  Compliance to diet, defined by the participants' persistence in low protein diet, by outpatient follow-up and telephone follow-up.
Nutritional status | 1 year
  Nutritional status, evaluated by nutrition risk screening (NRS 2002), at the start and during the 1st year of investigators' intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Min Liu, M.D., Study Director — specify unaffiliated
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hu'nan, China

IPD SHARING:
Plan to Share IPD: Yes
During the experiment, investigators will share the development in the website.